CLINICAL TRIAL: NCT04758585
Title: Non-adherence to Pain Medication Increases Risk of Postoperative Frozen Shoulder: A Case Control Study
Brief Title: Non-adherence to Pain Medication Increases Risk of Postoperative Frozen Shoulder
Acronym: NaFS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kantonsspital Baden (Other)
Responsible Party: Principal Investigator, Richard Niehaus, Dr.med. Richard Niehaus, senior consultant of shoulder surgery, principle investigator, Kantonsspital Baden
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ID 2019-01392
Record Dates: First submitted 2021-02-11; First posted 2021-02-17 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Frozen Shoulder; Depression
MeSH Terms: conditions — Bursitis; Depression | interventions — Arthroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Active Comparator)
  Interventions: Procedure: Arthroscopy
- Control Group (No Intervention)

INTERVENTIONS:
Procedure: Arthroscopy — Shoulder Arthroscopy
  Arms: Study Group

SUMMARY:
Background: Postoperative Frozen-Shoulder (FS) or adhesive capsulitis is a relatively frequent complication (5-20%), even after simple arthroscopic shoulder surgeries. The pathophysiology is still unclear, but psychological factors may play a pivotal role. From clinical experience, the investigators hypothesized that participants, who are reluctant to take medications, particularly "pain-killers", have an increased incidence of postoperative FS. The investigators retrospectively compared participants with and without postoperative FS by their attitude towards medication and by depression scale questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Shoulder arthroscopy

Exclusion Criteria:

* Active frozen shoulder

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Self-developed questionnaire | 1 to 4 years postoperatively
  Adhereance to pain medication
PHQ 4 (Patient Health Questionnaire-4) | 1 to 4 years postoperatively
  Depression scale
SMS (Self-Medicating Scale) | 1 to 4 years postoperatively
  Patient's beliefs about self-medication

CONTACTS AND LOCATIONS:
Locations (1):
- Kantonsspital Baden, Baden, Canton of Aargau, Switzerland

IPD SHARING:
Plan to Share IPD: No